CLINICAL TRIAL: NCT07268339
Title: TRAIN - A Phase III Randomised Control Clinical Trial of Radiotherapy With Radiosensitisation Versus Intravesical Bacillus Calmette-Guerin Therapy for High-risk Non-muscle Invasive Bladder Cancer.
Brief Title: A Phase III Randomised Control Clinical Trial of Radiotherapy With Radiosensitisation Versus Intravesical Bacillus Calmette-Guerin Therapy for High-risk Non-muscle Invasive Bladder Cancer.
Acronym: TRAIN
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTsp223
Record Dates: First submitted 2025-09-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: High-Risk Non-Muscle Invasive Bladder Cancer
Keywords: non-muscle invasive bladder cancer; radiotherapy with radiosensitisation drugs; Bacillus Calmette-Guerin therapy
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm: BCG (Active Comparator): This arm is standard of care for this patient group. A standard protocol of 6 weekly intravesical installations, followed by 3 weekly instillations at approximately 3, 6, 12, 18, 24, 30 months and 36 months (depending on toxicity). Stock is taken and given per local hospital guildlines.
  Interventions: Other: BCG
- Experimental Arm: Radiotherapy with Radiosentiser drugs. (Experimental): Patients randomised to the radiotherapy arm will receive a hypofractionated schedule of external beam radiotherapy with a regimen of 55Gy in 20 fractions given once daily Monday to Friday over 4 weeks. Radiotherapy will be delivered with a conventional or 3D conformal technique with an empty bladder. It will be administered concurrently with a radiosensitiser (detailed below) selected by the treating physician according to local institutional practice.
  Radiosensitiser will be selected as one option from the following:
  * Gemcitabine 75-100mg/m2 administered once a week during a four-week radiotherapy course. Cycle 1 will be given on the first radiotherapy day, to a planned total of 4 cycles. 2-4 hours prior to radiotherapy
  * 5-FU and Mitomycin C - Fluorouracil 500mg/m2 Days 1-5 and 16-20 via continuous infusion. Mitomycin C 12mg/m2 Day 1 via intravenous infusion
  * Carbogen and nicotinamide (CON) - 2% CO2 and 98% O2 Carbogen will be delivered through a closed breathing system with
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — Radiotherapy - 55Gy in 20 fractions treating once daily Monday to Friday over 4 weeks.
  Arms: Experimental Arm: Radiotherapy with Radiosentiser drugs.
Other: BCG — BCG protocol of 6 weekly intravesical instillations, followed by 3 weekly instillations at 3, 6, 12, 18, 24, 30, 36 months.
  Arms: Control Arm: BCG

SUMMARY:
In the UK 20,000 people develop urothelial bladder cancer each year with 75-80% having Non-Muscle Invasive Bladder Cancer (NMIBC). The current standard of care for patients with High Risk-NMIBC (HR-NMIBC) is either surgery to remove the tumour (transurethral resection of bladder tumour; TURBT) followed by BCG (Bacillus Calmette Guérin, an immunotherapy drug) given directly into the bladder, or surgery to remove the bladder (cystectomy). BCG is given weekly for six weeks followed by maintenance treatment up to 3 years. However, in up to 50% of patients their cancer returns (recurrence) or gets worse (progression) after BCG and 25% stop treatment due to side effects. Globally BCG supply has been restricted in recent years has increased HR-NMIBC recurrence rates and costs. Improved treatments are required, to prevent recurrence, progression and cystectomy, and mitigate the effects of unpredictable supply.

Trimodality treatment (TMT) is maximal TURBT + radiotherapy + a radiosensitiser (gemcitabine, mitomycin C/fluorouracil or carbogen/nicotinamide) and is an equivalent alternative treatment to cystectomy for muscle-invasive bladder cancer (MIBC). TMT is not routinely used for HR-NMIBC. A study found that 54% of HR-NMIBC patients who received TMT did not have recurrence within 5 years. Modern radiotherapy is expected to further improve outcomes and minimise side-effects.

Patients will be randomised 1:1 to BCG or radiotherapy with radiosensitisation. Patients randomised to the experimental arm will receive 55Gy in 20 fractions. Investigators can then choose from three different options for the radiosensitiser. TRAIN will test if radiotherapy with radiosensitisation improves outcomes for people with HR-NMIBC compared to BCG.

TRAIN will recruit 328 patients with HR-NMIBC following maximal TURBT. All patients will be followed up for a minimum of two years to record their response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with histologically confirmed grade 3 T1 N0 M0 transitional cell carcinoma, OR carcinoma in situ of the bladder (and N0 M0), OR both, with detrusor muscle present in the biopsy specimen if T1 disease (or a repeat resection that does contain muscle that is clear)
* Suitable for BCG treatment
* Suitable for radiotherapy and radiosensitisation according to the schedule of administration outlined in the Radiotherapy Planning Guidance document.
* Life expectancy over 12 months
* ECOG performance status 0 - 2
* Age >=16 years
* Provided written informed consent

Exclusion Criteria:

* MDT selected patients with HR-NMIBC who are deemed best suited for primary cystectomy (patients that have had this treatment recommendation but then decline cystectomy remain eligible for TRAIN)
* Previous radiotherapy to the pelvis
* Previous intravesical therapy
* Poor bladder function (IPSS >16)
* A recent or current other cancer. Current non-melanoma skin cancer, cervical carcinoma in situ or localized prostate cancer not requiring current treatment are permissible, as is a history of a separate other malignancy having completed all active treatment ≥2 years previously and without evidence of relapse
* Pre-existing medical conditions that preclude treatment options in either trial arm
* Patient currently recruited to another interventional trial or participation within an interventional clinical trial within 3 months of the point of registration within TRAIN.
* Pregnant or breast-feeding
* Not able to use appropriate adequate effective contraception during and for 3 months after the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2031-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
To compare event-free survival between BCG and radiotherapy with radiosensitisation. | From baseline to at least 96 weeks after initial of treatment.
  Event-free survival is defined as recurrence of CIS or high-risk non-muscle invasive papillary tumour, continued presence of HR NMIBC even after treatment completion, progression to muscle-invasive disease, distant metastatic bladder cancer, cystectomy (for any reason) or death from any cause.

SECONDARY OUTCOMES:
To determine the difference between BCG and radiotherapy in terms of patient-reported symptoms. | From baseline to at least 96 weeks post treatment.
  Patient-reported outcomes will be assessed via questionnaires, including the RTOG (late bladder and intestinal toxicity) questionnaire.
To evaluate each component of the primary outcome comparing between BCG and radiotherapy with radiosensitisation. | From baseline to at least 96 weeks post treatment.
  The following event outcomes will be analyzed using the Cox proportional hazards model to estimate hazard ratios, and Kaplan-Meier analysis will be used to estimate event rates.
  * Recurrence-free survival (RFS) defined as time from randomisation to recurrence of non-muscle invasive papillary tumour. Patients are censored at the last follow-up if event free.
  * Progression-free survival (PFS) defined as time from randomisation to progression to muscle-invasive disease. Patients are censored at the last follow-up if event free.
  * Metastasis-free survival (MFS) defined as time from randomisation to progression to distant metastatic bladder cancer. Patients are censored at the last follow-up if event free.
  * Cystectomy-free survival (CFS) defined as time from randomisation to cystectomy. Patients are censored at the last follow-up if event free
  * Overall survival (OS) defined as time from randomisation to death due to any cause. Patients are censored at the last follow-up if event free
To establish the tolerability and safety of radiotherapy. | From baseline to at least end of 4 week treatment.
  MedDRA coded adverse events graded using CTCAE v5.0.
To determine the difference in cancer specific survival between groups. | From baseline to at least 96 weeks post treatment.
  Cancer specific survival defined as time from randomisation to death from cancer. Patients who die of a cause other than the cancer under study or who are lost to follow-up are censored at death or the last date on which they were known to be alive.
To determine the difference in treatment fidelity between the groups. | From baseline to at least 96 weeks post treatment.
  Treatment fidelity defined as how well each group implemented treatment as intended. Summary statistics will be presented for any treatment delays, missed treatment, those not starting treatment, and those who completed treatment, by group.
To determine the cost-effectiveness of radiotherapy with radiosensitisation compared to BCG. | From Baseline to at least 96 weeks post treatment.
  * Within trial analysis. Total costs and QALYs for radiotherapy with radiosensitisation compared to BCG during the trial period.
  * Economic modelling. Total costs and QALYs for radiotherapy with radiosensitisation compared to BCG extrapolated beyond the trial period.
To determine the difference between BCG and radiotherapy in terms of patient-reported symptoms. | From baseline to at least 96 weeks post treatment.
  Patient-reported outcomes will be assessed via questionnaires, including the EQ-5D questionnaire.
To determine the difference between BCG and radiotherapy in terms of patient-reported symptoms. | From baseline to at least 96 weeks post treatment.
  Patient-reported outcomes will be assessed via questionnaires, including the IPSS questionnaire.
To determine the difference between BCG and radiotherapy in terms of patient-reported symptoms. | From baseline to at least 96 weeks post treatment.
  Patient-reported outcomes will be assessed via questionnaires, including the QLQ-C30 questionnaire.
To determine the difference between BCG and radiotherapy in terms of patient-reported symptoms. | From baseline to at least 96 weeks post treatment.
  Patient-reported outcomes will be assessed via questionnaires, including the QLQ-NMIBC24 questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available, including data dictionaries, for approved data-sharing requests. Individual participant data will be shared that underlie the results reported in this article, after de-identification and normalisation of information (text, tables, figures, and appendices). The study protocol and statistical analysis plan will also be available.
Supporting Information: Study Protocol, SAP
Time Frame: Anonymous data will be available for request from three months after publication of the article, to researchers who provide a completed Data Sharing request form that describes a methodologically sound proposal, for the purpose of the approved proposal and if appropriate, signed a Data Sharing Agreement.
Access Criteria: Data will be shared once all parties have signed relevant data-sharing documentation, covering SCTU conditions for sharing and if required, an additional Data Sharing Agreement from Sponsor. Proposals should be directed to ctu@soton.ac.uk.
URL: https://www.southampton.ac.uk/research/institutes-centres/clinical-trials-unit/working-with-us#:~:text=Data%20access%20is%20administered%20through%20the%20SCTU%20Data,form%202.%20email%20the%20completed%20form%20to%20ctuadmin%40soton.ac.uk

REFERENCES:
- See also: The TRAIN trial website. — https://www.southampton.ac.uk/ctu/train.page